CLINICAL TRIAL: NCT05454163
Title: Evaluation of Chronic Rhinosinusitis in Children Managed for Cervicofacial Mesenchymal Malignancy
Brief Title: Post-radiotherapy Rhinosinusitis in Children
Acronym: PRRSC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0549; 2022-A00422-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Cancer; Chronic Sinusitis
Keywords: Post-treatment chronic sinusitis; Pediatric cancer; Sinusitis; Quality of life
MeSH Terms: conditions — Neoplasms; Sinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed patients
  Interventions: Other: SNOT 22 questionnaire
- Non exposed patients

INTERVENTIONS:
Other: SNOT 22 questionnaire — 22 items, score between 0 and 5; sum, minimum = 0, maximum = 110; higher score = higher impact on quality of life)
  Groups: Exposed patients

SUMMARY:
Chronic rhinosinusitis (CRS) is a frequent complication of facial cancer treatment, mainly related to radiotherapy. However, while radiological involvement is frequent, clinical expression seems less important.

Few studies have investigated the incidence of this condition in the pediatric population while its evolution seems to be very chronic even if a partial improvement may occur with time.

Our objective is therefore to study the impact of CSR in children treated for cancer of the cervicofacial region, to evaluate its incidence and medium-term evolution in order to determine whether it is necessary to set up a specific follow-up in these patients.

The clinical impact of CSR is assessed by a specific SNOT 22 questionnaire in children treated for a head-neck mesenchymal malignancy in comparison with a control population consisting of children treated for a mesenchymal malignancy of non-head-neck location.

ELIGIBILITY:
Inclusion Criteria:

* Study population: all patients under 18 years of age managed for a head neck mesenchymal cancer between January 1, 2018 and December 31, 2024
* Control population: all patient under 1 years of age managed for non -head neck mesenchymal cancer between January 1, 2018 and December 31, 2024

Exclusion Criteria:

* Patients with hematological tumors;
* Patients with mucociliary pathologies or proven allergic rhinitis before the diagnosis of cancer
* Patients who have required surgical treatment that has removed more than half of the sinus cavities
* Tumor recurrence at the time of inclusion
* Sinus surgery between the last radiological check-up and inclusion
* Administrative reasons: inability to receive informed information.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population (called exposed) concerns all patients under 18 years of age managed for a head neck mesenchymal cancer between January 1, 2018 and December 31, 2024 in the pediatric surgery department of the Lille University Hospital.
  The control population (called non-exposed) included children treated during the same period for a non-head neck mesenchymal malignant cancer
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Impact of CRS in pediatric patients by Sino-Nasal Outcome Test-22 (SNOT 22) | >1 year to <4 years after the end of oncologic treatment

SECONDARY OUTCOMES:
Incidence of CRS in pediatric patients after head neck mesenchymal cancer management | 1 year after the end of the oncologic treatment
Correlation between SNOT 22 and clinical assessment by PADORES score | >1 year to <4 years after the end of oncologic treatment
Correlation between SNOT 22 and clinical assessment by lund-kennedy score | >1 year to <4 years after the end of oncologic treatment
Correlation between SNOT 22 and radiological assessment by Lund-Mackay score | >1 year to <4 years after the end of oncologic treatment
Radiological evolution of CRS by Lund-Mackay score | >1 year to <4 years after the end of oncologic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fayoux, MD,PhD, Principal Investigator — University Hospital, Lille